CLINICAL TRIAL: NCT01787227
Title: A Two Arm, Multi-Centre Clinical Evaluation of the NxTAG Respiratory Pathogen Panel (NxTAG RPP) in Patients With Clinical Signs and Symptoms of Respiratory Tract Infection
Brief Title: A Two Arm, Multi-Centre Clinical Evaluation of the NxTAG Respiratory Pathogen Panel
Status: Completed | Type: Observational
Sponsor: Luminex Molecular Diagnostics (Industry)
Responsible Party: Sponsor
Other Study IDs: TDP-736-272
Record Dates: First submitted 2013-02-01; First posted 2013-02-08 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-03

CONDITIONS: Respiratory Tract Infection; Bronchitis; Bronchiolitis; Pneumonia
MeSH Terms: conditions — Respiratory Tract Infections; Bronchitis; Bronchiolitis; Pneumonia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Nasopharyngeal swab
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Blinded, Pre-selected Arm: For targets that exhibit lower prevalence rates in the intended use population, banked, pre-selected, positive clinical specimens will be tested.
  Interventions: Device: xTAG RPP
- Blinded, Prospective Arm: Diagnostic accuracy for the more prevalent targets will be evaluated in prospectively collected, de-identified, left-over, clinical specimens accrued during the 2012/2013 flu season.
  Interventions: Device: xTAG RPP

INTERVENTIONS:
Device: xTAG RPP

SUMMARY:
xTAG RPP assay is a PCR-based assay to detect the presence or absence of viral and bacterial DNA / RNA in clinical specimens (nasopharyngeal swabs).

The objective of this study is to establish diagnostic accuracy of the xTAG RPP.

ELIGIBILITY:
Inclusion Criteria:

* The specimen is a nasopharyngeal swab.
* The specimen is from a pediatric or adult, male or female subject who is either hospitalized, admitted to a hospital emergency department, visiting an outpatient clinic or resident of a long-term care facility.
* The specimen is from a patient exhibiting clinical signs and symptoms of respiratory tract infection such as fever, sore throat, shortness of breath, bronchitis, bronchiolitis and pneumonia.

Exclusion Criteria:

* The specimen is not a nasopharyngeal swab.
* The specimen is from an individual who does not exhibit clinical signs and symptoms of respiratory tract infection.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Clinical specimens collected from patients with clinical signs and symptoms of respiratory tract infection who are either hospitalized, admitted to emergency departments or visiting outpatient clinics.
Sampling Method: Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2015-01; Primary Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy will be expressed in terms of clinical sensitivity and specificity for each claimed target. | Within the first year after sample extraction
  Accuracy determinations (diagnostic sensitivity and specificity, positive and negative agreement) were based on the fraction of comparator positive (or negative) results which were also positive (or negative) by xTAG RPP.

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Liu, Ph.D, Study Director — Luminex Molecular Diagnostics; James Mahony, Ph.D, FCCM, FAAM, Principal Investigator — St. Joseph's Health Care London; Richard Buller, PhD, D (ABMM), Principal Investigator — St. Louis Children's Hospital; Arundhati Rao, M.D., Ph.D., Principal Investigator — Scott and White Hospital & Clinic; Christine Ginocchio, Ph.D., M.T.(A.S.C.P.), Principal Investigator — North Shore-LIJ Health System Laboratories, NY
Locations (4):
- United States (3):
  - St. Louis Children's Hospital, St Louis, Missouri
  - North Shore-LIJ Health System Laboratories, Lake Success, New York
  - Scott and White Memorial Hospital, Temple, Texas
- St. Joseph's Hospital, Hamilton, Ontario, Canada